CLINICAL TRIAL: NCT05526456
Title: Department of Thoracic Surgery, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Brief Title: Mapping of Lymph Node Metastasis and Survival For pN+ Superficial Esophageal Squamous Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: National Cancer Center, China (Other)
Responsible Party: Principal Investigator, Yin Li, Department of Thoracic Surgery, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, National Cancer Center, China
Other Study IDs: 20/388-2584
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: National Cancer Center/Cancer Hospital
MeSH Terms: interventions — Esophagectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Esophagectomy — McKeown, Ivor-Lewis, and Sweet procedure

SUMMARY:
With the deeper tumor invasion, the higher LNM rate beside the bilateral recurrent laryngeal nerves(RLN) was.

ELIGIBILITY:
Inclusion Criteria:

* Our predefined search strategy identified pT1N+ ESCC cases without preoperative treatment, between February 2012 and April 2022.

Exclusion Criteria:

* The patients were excluded because they were (1)less than 10 lymph nodes removed; (2) lacked specific sites of LNM; or (3) incomplete follow-up information.

Ages: 44 Years to 73 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Among the 207 patients, 22 were in the T1a stage, whereas 185 were in the T1b stage. The invasion depth was EP in 2, LPM in 1, MM in 17, SM1 in 37, SM2 in 39 and SM3 in 97 patients
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
LNM rates of the 207 thoracic T1N+ ESCC patients. | 2012.2-2022.4